CLINICAL TRIAL: NCT03084055
Title: A Pilot Randomized Controlled Trial of a Web-based Intervention Using Behavioral Activation and Physical Activity for Adults With Depression: the eMotion Study.
Brief Title: A Pilot Randomized Controlled Trial of an Intervention for Adults With Depression: the eMotion Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1516/029
Record Dates: First submitted 2016-06-15; First posted 2017-03-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- eMotion intervention (Experimental): Subjects randomised to the intervention arm will receive eMotion for two months. eMotion is comprised of a series of weekly audio visual modules designed to increase exposure to positive activities and physical activity.
  Interventions: Behavioral: eMotion
- Waiting list control (No Intervention): Subjects in the waiting list control group will be given no intervention for two months; the control group will then be able to access eMotion if they wish but this will not form part of the research project

INTERVENTIONS:
Behavioral: eMotion — eMotion is comprised of a series of weekly audio visual modules designed to increase exposure to positive activities and physical activity
  Arms: eMotion intervention

SUMMARY:
Physical activity has many potential mood enhancing benefits, and may be as effective as anti-depressants and psychological therapies for treating depression and low mood. However, getting people with depression to become more active is challenging. Behavioural Activation (BA) is an evidenced based psychotherapeutic treatment that focuses on increasing exposure to positive environmental stimuli which could provide an effective delivery mechanism for increasing physical activity for people who are more sedentary than the general population. The purpose of this study is to examine the feasibility of delivering a theory informed online intervention combining physical activity and BA (eMotion) to people with depression, and to examine its effects on depressive symptoms and physical activity.

DETAILED DESCRIPTION:
A randomised controlled trial (RCT) design will be used in this study. 120 participants experiencing depressive symptoms (>10 on the PHQ-8) over the age of 18 will be recruited from the community. Participants will be eligible to participate if the over 18, score over 10 on the PHQ-8 and, are able to walk unaided for at least 5 minutes and have access to the internet. Following baseline measures, participants will be randomised in a 1:1 ratio to the intervention or waiting list control arm and be followed up at 2 and 5 months. Those randomised to the intervention arm will receive eMotion which is comprised of a series of weekly audio visual modules designed to increase exposure to positive activities and physical activity. Main outcomes of interest include recruitment, retention, fidelity and acceptability. Baseline and follow up measures will also include the PHQ-8, and objective (GENEActvie accelerometers) and subjective (IPAQ) measures of physical activity. A parallel process evaluation will run alongside the RCT.

If effective, this intervention has the potential to improve depressive symptoms in a wide range of hard to reach people in the community and increase their physical activity. Further evaluation in a full scale RCT is planned pending results of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged ≥18 years).
* Adults with possible mild to moderately severe depression reflected by a score of between 10 and 23 (i.e. moderate to moderately severe depressive symptoms) on the Patient Health Questionnaire (PHQ-8) as has been done in previous studies looking at low mood and depressive symptoms.
* Adults living in the UK.
* Having access to the internet.
* Able to walk continuously and unaided for a minimum of 5 minutes.
* Provision of informed consent to participate.

Exclusion Criteria:

* Adults (aged <18 years).
* Adults without possible mild to moderately severe depression reflected by a score of between 10 and 23 (i.e. moderate to moderately severe depressive symptoms) on the Patient Health Questionnaire (PHQ-8) as has been done in previous studies looking at low mood and depressive symptoms.
* Adults not living in the UK.
* No access to the internet.
* Not able to walk continuously and unaided for a minimum of 5 minutes.
* Lacking capacity to give informed consent to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
Depression | Two months
  Depression will be measured using tThe Personal Health Questionnaire (PHQ-8). The PHQ-8 is an 8 item measure used to measure the frequency of depressive symptoms. This is a freely available brief self-report questionnaire which assesses depressive symptoms based on the Diagnostic and Statistical Manual for Mental Disorders (DSM-IV). Each item is rated on a scale of 0 to 3 with a maximum score of 24. It has been shown to have good validity, reliability, sensitivity and specificity. It has also been shown to discriminate between levels of major and major severe depression being 10-19, and 20-23 respectively (Kroenke et al., 2009)

SECONDARY OUTCOMES:
Objective Physical Activity | Two months
  Objective physical activity will be assessed using GeneACTIVE wrist worn accelerometers. The accelerometer is a small wrist worn device that measures and records acceleration. 1 minute epochs will be used to measure movement, with higher counts per minute reflecting higher levels of physical activity as recommended in previous studies (Helgadóttir, Forsell, & Ekblom, 2015; Mailey et al., 2010).
Anxiety | Two months
  General Anxiety Disorder (GAD-7) is a 7 item scale which measures symptoms and severity of anxiety based on the DSM-IV criteria and included in the minimum IAPT data set (Spitzer, Kroenke, Williams, & Lowe, 2006).
Affective Mood State | Two months
  Ecological Momentary Assessment of Mood (EMA) will be taken using a one item 10 point scale asking the participant to rate their mood where 1 = sad and 10 = happy. This will be taken twice per day randomly over five days during baseline data collection and at two months follow up using 'Text local', a text messaging service which allows participants to respond with a number response indicating their current mood at that point in time. This approach is adapted from previous research (van Rijsbergen, Bockting, Berking, Koeter, & Schene, 2012).
Self-reported physical activity | Two months
  Self-reported physical activity will be measured using the short-form IPAQ which measures Minutes per week of moderate to vigorous physical activity will be assessed by using the International Physical Activity Questionnaire (IPAQ). The IPAQ is a valid cross national measure of self-reported physical activity (Craig et al., 2003).

OTHER OUTCOMES:
Fidelity of receipt | Two months
  The website will be assessed by asking questions understanding, perceived understanding the key learning goals for participants in all groups.
Fidelity of enactment | Two months
  Fidelity of enactment will be measured by asking participants in all groups if they have carried out specific behaviour change techniques relating to physical activity, and behavioural activation along with rating confidence.
Participant satisfaction | Two months
  The Client Satisfaction Questionnaire - Short Form (CSQ-SF). This is a 4 item measure which will be used to assess participant satisfaction in eMotion 2 months post randomization.
Participant views of intervention | Two months
  Qualitative interviews after the final intervention session, all participants who receive eMotion will be invited to participate in a semi structured interview over the phone. The purpose of this is to further examine the acceptability of the intervention and any suggestions for improvement which can be absorbed into a next trial.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Lambert, MSc, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lambert JD, Greaves CJ, Farrand P, Price L, Haase AM, Taylor AH. Web-Based Intervention Using Behavioral Activation and Physical Activity for Adults With Depression (The eMotion Study): Pilot Randomized Controlled Trial. J Med Internet Res. 2018 Jul 16;20(7):e10112. doi: 10.2196/10112. PMID 30012547